CLINICAL TRIAL: NCT03933449
Title: A Phase III Randomized Open-Label Study of Single Agent Pembrolizumab vs Physicians' Choice of Single Agent Docetaxel, Paclitaxel, or Irinotecan in Subjects With Advanced/Metastatic Adenocarcinoma and Squamous Cell Carcinoma of the Esophagus That Have Progressed After First-Line Standard Therapy (KEYNOTE-181)
Brief Title: Study of Pembrolizumab (MK-3475) Versus Investigator's Choice of Chemotherapy for Participants With Advanced Esophageal/Esophagogastric Junction Carcinoma That Progressed After First-Line Therapy (MK-3475-181/KEYNOTE-181)-China Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-181 China Extension; 163145 (Registry Identifier: JAPAN-CTI); MK-3475-181 (Other: Merck); KEYNOTE-181 (Other: Merck)
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Results first posted 2020-02-26 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Esophageal Carcinoma; Esophagogastric Junction Carcinoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Programmed Death-Ligand 2 (PDL2, PD-L2); Gene expression profiling (GEP)
MeSH Terms: conditions — Esophageal Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Paclitaxel; Docetaxel; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab (Experimental): Participants receive pembrolizumab 200 mg intravenously (IV) on Day 1 of every 21-day (3-week) cycle for up to 35 administrations (up to ~2 years). Participants who complete the first course of up to 35 administrations of pembrolizumab (~2 years) but progress after discontinuation, may be eligible for a second course of pembrolizumab at the investigator's discretion, at the same dose and schedule at 200 mg IV on Day 1 of each 3-week cycle for up to 17 cycles (up to ~1 year).
  Interventions: Biological: pembrolizumab
- Chemotherapy (Active Comparator): Participants receive Investigator's choice of chemotherapy: paclitaxel 80-100 mg/m^2 IV on Days 1, 8, and 15 of every 28-day (4-week) cycle, OR docetaxel 75 mg/m^2 IV on Day 1 of every 21-day (3-week) cycle, OR irinotecan 180 mg/m^2 IV on Day 1 of every 14-day (2-week) cycle (up to ~2 years).
  Interventions: Drug: paclitaxel; Drug: docetaxel; Drug: irinotecan

INTERVENTIONS:
Biological: pembrolizumab — IV infusion
  Other Names: KEYTRUDA®; MK-3475
  Arms: Pembrolizumab
Drug: paclitaxel — IV infusion
  Other Names: TAXOL®
  Arms: Chemotherapy
Drug: docetaxel — IV infusion
  Other Names: TAXOTERE®
  Arms: Chemotherapy
Drug: irinotecan — IV infusion
  Other Names: CAMPTOSAR®
  Arms: Chemotherapy

SUMMARY:
In the China extension study, Chinese participants with advanced or metastatic adenocarcinoma or squamous cell carcinoma of the esophagus or Siewert type I adenocarcinoma of the esophagogastric junction (EGJ) that has progressed after first-line standard therapy will be randomized to receive either single agent pembrolizumab or the Investigator's choice of chemotherapy with paclitaxel, docetaxel, or irinotecan.

The primary extension study hypothesis is that treatment with pembrolizumab will prolong overall survival (OS) as compared to treatment with chemotherapy.

DETAILED DESCRIPTION:
The China extension study will include participants previously enrolled in China in the global study for MK-3475-181 (NCT02564263) plus those enrolled during the China extension enrollment period.

Per protocol, response/progression or adverse events during the second pembrolizumab course will not be counted towards efficacy outcome measures or safety outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-confirmed diagnosis of adenocarcinoma or squamous cell carcinoma of the esophagus or Siewert type I adenocarcinoma of the EGJ
* Metastatic disease or locally advanced, unresectable disease
* Life expectancy of greater than 3 months
* Measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
* Performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Documented radiographic or clinical disease progression on no more or less than one previous line of standard therapy
* Can provide either a newly obtained or archival tumor tissue sample for intra-tumoral immune-related testing and for anti-programmed cell death (PD)-1
* Participants of reproductive potential must be willing to use adequate contraception for the course of the study through 120 days after the last dose of pembrolizumab or through 180 days after the last dose of paclitaxel, docetaxel or irinotecan
* Adequate organ function

Exclusion Criteria:

* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of study medication
* Active autoimmune disease that has required systemic treatment in past 2 years
* Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study medication
* Known central nervous system (CNS) metastases and/or carcinomatous meningitis (includes past history or current metastasis)
* Has received prior anti-cancer monoclonal antibody (mAb), chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or not recovered from adverse events due to a previously administered agent
* Has had a severe hypersensitivity reaction to treatment with another mAb
* Prior therapy with a PD-1, anti-PD-Ligand 1 (PD-L1), or anti-PD-L2 agent, or previously participated in Merck pembrolizumab (MK-3475) study
* Has a known additional malignancy that has progressed or required active treatment within the last 5 years with the exception of curatively treated basal cell and squamous cell carcinoma of the skin and/or curatively resected in-situ cervical and/or breast cancers, and in-situ or intra-mucosal pharyngeal cancer
* Received a live vaccine within 30 days of the first dose of study medication
* Known history of Human Immunodeficiency Virus (HIV) infection
* Known history of or is positive for hepatitis B (hepatitis B surface antigen reactive) or known active hepatitis C [hepatitis C virus ribonucleic acid (RNA) or hepatitis C antibody is detected]
* History of non-infectious pneumonitis that required steroids or current pneumonitis
* Active infection requiring systemic therapy
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the study starting with the screening visit through 120 days after the last dose of pembrolizumab or through 180 days after the last dose of paclitaxel, docetaxel or irinotecan
* Known allergy, hypersensitivity, or contraindication to paclitaxel, docetaxel, or irinotecan or any components used in their preparation
* Experienced weight loss > 10% over ~2 months prior to first dose of study therapy
* Has ascites or pleural effusion by physical exam
* Has experienced documented objective radiographic or clinical disease progression during or after receiving more than 1 line of therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2022-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (23):
- China (23):
  - Anhui Provincial Hospital ( Site 0708), Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University ( Site 0707), Hefei, Anhui
  - Harbin Medical University Cancer Hospital ( Site 0714), Harbin, Heilongjiang
  - Wuhan Tongji Hospital ( Site 0724), Wuhan, Hubei
  - Hunan Cancer Hospital ( Site 0722), Changsha, Hunan
  - Jiangsu Cancer Hospital (Site 0704), Nanjing, Jiangsu
  - PLA Cancer Centre of Nanjing Bayi Hospital ( Site 0706), Nanjing, Jiangsu
  - Jilin Cancer Hospital ( Site 0718), Changchun, Jilin
  - The First Hospital Of Jilin University ( Site 0719), Changchun, Jilin
  - Zhejiang Cancer Hospital ( Site 0726), Hangzhou, Zhejiang
  - Beijing Cancer Hospital ( Site 0700), Beijing
  - Chinese PLA General Hospital (Site 0703), Beijing
  - Peking Union Medical College Hospital ( Site 0712), Beijing
  - Fujian Medical University Union Hospital ( Site 0721), Fuzhou
  - Fujian Province Cancer Hospital ( ( Site 0717), Fuzhou
  - The Second Affiliated Hospital of Zhejiang University School of Medicine ( Site 0705), Hangzhou
  - Sir Sun Sun Shaw Hosp, Zhejiang Univ,Oncology dept. ( Site 0720), Hangzhou
  - The Affiliated Hospital of Qingdao University ( Site 0709), Qingdao
  - Ruijin Hospital, Shanghai Jiaotong University ( Site 0701), Shanghai
  - Shanghai Chest Hospital ( Site 0727), Shanghai
  - Fudan University Shanghai Cancer Center ( Site 0723), Shanghai
  - Zhongshan Hospital affiliated to Fudan University ( Site 0715), Shanghai
  - Henan Cancer Hospital ( Site 0725), Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Cao Y, Qin S, Luo S, Li Z, Cheng Y, Fan Y, Sun Y, Yin X, Yuan X, Li W, Liu T, Hsu CH, Lin X, Kim SB, Kojima T, Zhang J, Lee SH, Bai Y, Muro K, Doi T, Bai C, Gu K, Pan HM, Bai L, Yang JW, Cui Y, Lu W, Chen J. Pembrolizumab versus chemotherapy for patients with esophageal squamous cell carcinoma enrolled in the randomized KEYNOTE-181 trial in Asia. ESMO Open. 2022 Feb;7(1):100341. doi: 10.1016/j.esmoop.2021.100341. Epub 2021 Dec 29. PMID 34973513
- See also: Merck Oncology Clinical Trial Information — http://merckoncologyclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, response/progression or adverse events during the second pembrolizumab course were not counted towards efficacy outcome measures or safety outcome measures.
  Final analysis of all outcome measures was done at the protocol-specified analysis cutoff of 13-Feb-2019.
Groups:
- Pembrolizumab: Participants received pembrolizumab 200 mg intravenously (IV) on Day 1 of every 21-day (3 week) cycle for up to 35 administrations (up to ~2 years). Participants who completed the first course of up to 35 administrations of pembrolizumab (~2 years) but progressed after discontinuation, were eligible for a second course of pembrolizumab at the investigator's discretion, at the same dose and schedule at 200 mg IV on Day 1 of each 3-week cycle for up to 17 cycles (up to ~1 year).
- Chemotherapy: Participants received Investigator's choice of chemotherapy for up to ~2 years: paclitaxel 80-100 mg/m^2 IV on Days 1, 8, and 15 of every 28-day (4-week) cycle, OR docetaxel 75 mg/m^2 IV on Day 1 of every 21-day (3-week) cycle, OR irinotecan 180 mg/m^2 IV on Day 1 of every 14-day (2-week) cycle.
Period: Overall Study
Arm/Group | Pembrolizumab | Chemotherapy
Started | 62 | 61
Treated | 62 | 59
Received Second Course | 1 | 0
Discontinued | 62 | 61
Completed | 0 | 0
Not Completed | 62 | 61
Not completed — Adverse Event | 6 | 4
Not completed — Death | 55 | 57
Not completed — Sponsor Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab | Chemotherapy | Total
Number analyzed (Participants) | 62 | 61 | 123
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.1 (7.0) | 59.6 (7.0) | 59.9 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 57 | 58 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 62 | 61 | 123
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 62 | 61 | 123
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Programmed Death-Ligand 1 (PD-L1) Status: Combined Positive Score (CPS) [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression levels by immunohistochemistry assay on tumor tissue from a newly obtained biopsy. PD-L1 CPS was calculated as the number of PD-L1 positive cells (tumor cells, macrophages, lymphocytes) divided by the total tumor cells and is expressed as a percentage. Participants were classified based on their PD-L1 tumor status as being either PD-L1 CPS ≥10 or PD-L1 CPS <10.
  Participants
    PD-L1 CPS ≥10 | 25 | 29 | 54
    PD-L1 CPS <10 | 35 | 31 | 66
    Not Evaluable | 2 | 1 | 3
Tumor Histology [Count of Participants; unit: Participants] — Participants were classified based on their tumor histology (cell type) as either having squamous cell carcinoma or having adenocarcinoma of esophagus and esophagogastric junction (EGJ) Siewert type I.
  Participants
    Squamous cell carcinoma | 60 | 59 | 119
    Adenocarcinoma of esophagus & EGJ Siewert type I | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in All Participants
Description: OS was defined as the time from randomization to death due to any cause. Median OS for the first pembrolizumab course in all participants is presented.
Time Frame: From randomization through final analysis data cutoff date of 13-Feb-2019 (Up to ~24 months)
Population: The efficacy analysis population consisted of all randomized participants. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Pembrolizumab: Participants received pembrolizumab 200 mg intravenously (IV) on Day 1 of every 21-day (3 week) cycle for up to 35 administrations (up to ~2 years).
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 62 | 61
Months | 8.4 [5.8 to 10.9] | 5.6 [4.5 to 7.3]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.0015, Log Rank — One-sided p-value based on log-rank test; Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.36 to 0.82] — Based on Cox regression model with treatment as a covariate

2. Primary Outcome: Overall Survival (OS) in Participants With Programmed Death-Ligand 1 Combined Positive Score ≥10 (PD-L1 CPS ≥10)
Description: OS was defined as the time from randomization to death due to any cause. Median OS for the first pembrolizumab course in participants with a PD-L1 CPS ≥10 is presented.
Time Frame: From randomization through final analysis data cutoff date of 13-Feb-2019 (Up to ~24 months)
Population: The efficacy analysis population consisted of all randomized participants with a PD-L1 CPS ≥10. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 25 | 29
Months | 12.0 [6.6 to NA] — NA=OS Upper Limit could not be calculated due to an insufficient number of deaths on study as of the data cutoff date of 13-Feb-2019 | 5.3 [4.1 to 8.2]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.0008, Log Rank — One-sided p-value based on log-rank test; Hazard Ratio (HR) = 0.34, 95% CI 2-sided [0.17 to 0.69] — Based on Cox regression model with treatment as a covariate

3. Primary Outcome: Overall Survival (OS) in Participants With Squamous Cell Carcinoma (SCC) of the Esophagus
Description: OS was defined as the time from randomization to death due to any cause. Median OS for the first pembrolizumab course in participants with SCC of the esophagus is presented.
Time Frame: From randomization through final analysis data cutoff date of 13-Feb-2019 (Up to ~24 months)
Population: The efficacy analysis population consisted of all randomized participants with SCC of the esophagus. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 60 | 59
Months | 8.4 [5.8 to 10.9] | 5.6 [4.5 to 7.3]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.0021, Log Rank — One-sided p-value based on log-rank test; Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.37 to 0.83] — Based on Cox regression model with treatment as a covariate

4. Secondary Outcome: Objective Response Rate (ORR) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in All Participants
Description: ORR was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) as assessed using RECIST 1.1 by central imaging vendor review. The percentage of all participants who experienced a CR or PR for the first pembrolizumab course is presented.
Time Frame: From randomization through final analysis data cutoff date of 13-Feb-2019 (Up to ~24 months)
Population: The efficacy analysis population consisted of all randomized participants who experienced a confirmed response (CR or PR). Participants were included in the treatment group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 62 | 61
Percentage of Participants | 16.1 [8.0 to 27.7] | 3.3 [0.4 to 11.3]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.0084, Miettinen & Nurminen method — One-sided p-value for testing. H0: difference in %=0 versus H1: difference in %>0; Difference in Percentages = 12.9, 95% CI 2-sided [2.7 to 24.5]

5. Secondary Outcome: Objective Response Rate (ORR) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Participants With Programmed Death-Ligand 1 Combined Positive Score ≥10 (PD-L1 CPS ≥10)
Description: ORR was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) as assessed using RECIST 1.1 by central imaging vendor review. The percentage of participants with a PD-L1 CPS ≥10 who experienced a CR or PR for the first pembrolizumab course is presented.
Time Frame: From randomization through final analysis data cutoff date of 13-Feb-2019 (Up to ~24 months)
Population: The efficacy analysis population consisted of all randomized participants with a PD-L1 CPS ≥10 who experienced a confirmed response (CR or PR). Participants were included in the treatment group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 25 | 29
Percentage of Participants | 24.0 [9.4 to 45.1] | 6.9 [0.8 to 22.8]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.0403, Miettinen & Nurminen method — One-sided p-value for testing. H0: difference in %=0 versus H1: difference in %>0; Difference in Percentages = 17.1, 95% CI 2-sided [-2.3 to 38.0]

6. Secondary Outcome: Objective Response Rate (ORR) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Participants With Squamous Cell Carcinoma (SCC) of the Esophagus
Description: ORR was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) as assessed using RECIST 1.1 by central imaging vendor review. The percentage of participants with SCC of the esophagus who experienced a CR or PR for the first pembrolizumab course is presented.
Time Frame: From randomization through final analysis data cutoff date of 13-Feb-2019 (Up to ~24 months)
Population: The efficacy analysis population consisted of all randomized participants with SCC of the esophagus who experienced a confirmed response (CR or PR). Participants were included in the treatment group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 60 | 59
Percentage of Participants | 16.7 [8.3 to 28.5] | 3.4 [0.4 to 11.7]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.0083, Miettinen & Nurminen method — One-sided p-value for testing. H0: difference in %=0 versus H1: difference in %>0; Difference in Percentages = 13.3, 95% CI 2-sided [2.8 to 25.2]

7. Secondary Outcome: Progression-free Survival (PFS) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in All Participants
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of ≥1 new lesions was also considered PD. Median PFS for the first pembrolizumab course as assessed by central imaging vendor review per RECIST 1.1 in all participants is presented.
Time Frame: From randomization through final analysis data cutoff date of 13-Feb-2019 (Up to ~24 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 62 | 61
Months | 2.5 [2.1 to 4.1] | 2.8 [2.0 to 4.2]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.177, Log Rank — One-sided p-value based on log-rank test; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.58 to 1.23] — Based on Cox regression model with treatment as a covariate

8. Secondary Outcome: Progression-free Survival (PFS) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Participants With Programmed Death-Ligand 1 Combined Positive Score ≥10 (PD-L1 CPS ≥10)
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of ≥1 new lesions was also considered PD. Median PFS for the first pembrolizumab course as assessed by central imaging vendor review per RECIST 1.1 is presented for participants with a PD-L1 CPS ≥10.
Time Frame: From randomization through final analysis data cutoff date of 13-Feb-2019 (Up to ~24 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 25 | 29
Months | 4.0 [2.1 to 6.1] | 4.0 [2.0 to 5.3]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.238, Log Rank — One-sided p-value based on log-rank test; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.44 to 1.46] — Based on Cox regression model with treatment as a covariate

9. Secondary Outcome: Progression-free Survival (PFS) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Participants With Squamous Cell Carcinoma (SCC) of the Esophagus
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of ≥1 new lesions was also considered PD. Median PFS for the first pembrolizumab course as assessed by central imaging vendor review per RECIST 1.1 is presented for participants with SCC of the esophagus.
Time Frame: From randomization through final analysis data cutoff date of 13-Feb-2019 (Up to ~24 months)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 60 | 59
Months | 2.3 [2.1 to 4.1] | 2.8 [2.0 to 4.2]
Statistical Analysis 1: Comparison: Pembrolizumab vs Chemotherapy; Test type: Superiority; p = 0.171, Log Rank — One-sided p-value based on log-rank test; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.57 to 1.23] — Based on Cox regression model with treatment as a covariate

10. Secondary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. The number of participants who experienced ≥1 AE for the first pembrolizumab course are presented.
Time Frame: From randomization through final analysis data cutoff date of 13-Feb-2019 (Up to ~24 months)
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 62 | 59
Participants | 62 | 56

11. Secondary Outcome: Number of Participants Discontinuing Study Treatment Due an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. The number of participants who discontinued study treatment due to an AE for the first pembrolizumab course are presented.
Time Frame: From randomization through final analysis data cutoff date of 13-Feb-2019 (Up to ~24 months)
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Chemotherapy
Number analyzed (Participants) | 62 | 59
Participants | 10 | 9

ADVERSE EVENTS:
Time Frame: From randomization through end-of-trial analysis data cutoff date of 14-March-2022 (Up to ~52 months)
Description: All-Cause Mortality (ACM): All randomized participants. Safety: All randomized participants who got ≥1 dose of study treatment.
  Per protocol, disease progression of cancer was not considered an AE unless related to study drug. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" unrelated to study drug are excluded as AEs.
  Participants who received a second course of pembrolizumab per protocol were monitored for ACM and AEs separately.
Groups:
- Pembrolizumab First Course: Participants received pembrolizumab 200 mg IV on Day 1 of every 21-day (3-week) cycle for up to 35 administrations (up to ~2 years).
- Pembrolizumab Second Course: Participants who completed the first course of up to 35 administrations of pembrolizumab (~2 years) but progressed after discontinuation, initiated a second course of pembrolizumab at the investigator's discretion, at the same dose and schedule at 200 mg IV on Day 1 of each 3-week cycle for up to 17 cycles (up to ~1 year).
Arm/Group | Pembrolizumab First Course | Chemotherapy | Pembrolizumab Second Course
All-Cause Mortality (participants affected / at risk) | 61/62 | 61/61 | 0/1
Serious Adverse Events (participants affected / at risk) | 23/62 | 23/59 | 0/1
Other Adverse Events (participants affected / at risk) | 58/62 | 55/59 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab First Course (N=62) | Chemotherapy (N=59) | Pembrolizumab Second Course (N=1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Oesophageal fistula (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 2 (2) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymph gland infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oesophageal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Anastomotic fistula (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acquired tracheo-oesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab First Course (N=62) | Chemotherapy (N=59) | Pembrolizumab Second Course (N=1)
Anaemia (Blood and lymphatic system disorders) | 19 (24) | 30 (49) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 7 (23) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 5 (17) | 0 (0)
Hypothyroidism (Endocrine disorders) | 12 (15) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 3 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 5 (7) | 4 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 10 (13) | 10 (14) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 17 (39) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 5 (5) | 3 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (8) | 6 (7) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (7) | 16 (22) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (8) | 19 (37) | 0 (0)
Asthenia (General disorders) | 12 (12) | 4 (4) | 0 (0)
Chest pain (General disorders) | 5 (6) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (6) | 10 (10) | 0 (0)
Malaise (General disorders) | 2 (2) | 6 (7) | 0 (0)
Pyrexia (General disorders) | 5 (8) | 9 (13) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 4 (4) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 9 (11) | 8 (8) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 11 (12) | 4 (6) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 6 (7) | 5 (8) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 4 (5) | 2 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 4 (6) | 2 (3) | 0 (0)
Blood chloride decreased (Investigations) | 0 (0) | 3 (4) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 3 (3) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 3 (3) | 4 (4) | 0 (0)
Blood urea increased (Investigations) | 2 (3) | 3 (4) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 8 (8) | 4 (4) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 8 (10) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (3) | 17 (55) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 3 (3) | 0 (0)
Platelet count decreased (Investigations) | 4 (4) | 5 (6) | 0 (0)
Tri-iodothyronine decreased (Investigations) | 1 (1) | 3 (3) | 0 (0)
Weight decreased (Investigations) | 13 (13) | 16 (18) | 0 (0)
White blood cell count decreased (Investigations) | 4 (7) | 28 (80) | 0 (0)
White blood cell count increased (Investigations) | 2 (2) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 11 (12) | 11 (13) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (6) | 3 (4) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 15 (24) | 11 (13) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 4 (7) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (5) | 11 (14) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 5 (7) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 3 (4) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (6) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 4 (4) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (3) | 3 (3) | 0 (0)
Proteinuria (Renal and urinary disorders) | 6 (6) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (20) | 7 (9) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (7) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT03933449/Prot_SAP_001.pdf